CLINICAL TRIAL: NCT05300490
Title: A Pilot Study of the Urinary Elimination Kinetics of Prednisolone After Intra-articular Injection in the Knee
Brief Title: Prednisolone Urinary Excretion Kinetics
Acronym: URIPRED
Status: Withdrawn | Type: Observational
Why Stopped: As practices had changed by the time this trial was being set up, there was no inclusion in this study.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8328
Record Dates: First submitted 2022-02-15; First posted 2022-03-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Articular Cartilage Disorder of Knee
Keywords: Doping; Prednisolone; Pharmacokinetics; Pharmacogenetics
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee infiltration: Patients requiring prednisolone knee infiltration as part of routine medical management
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — In this routine care study, all patients will receive a joint injection of prednisolone at a dose left to the discretion of the physician. The urinary excretion kinetics of this product and its metabolites will then be followed at different times. An association with metabolic genetic profile will be done.
  Other Names: Infiltration

SUMMARY:
The urinary elimination kinetics of glucocorticoids after intra-articular injection is very poorly documented. It is estimated that glucocorticoids may be present in the urine up to 6 weeks after intra-articular injection. However, this is not supported by any scientific literature. Despite this lack of evidence, in doping control practice, any presence of glucocorticoids in urine is accepted when the athlete provides evidence of an intra-articular injection that took place less than 6 weeks prior to the doping control. Many doping cases are open to challenge because they are based solely on measurements of prednisolone concentrations and its blood esterase product, prednisone. In order to demonstrate the use of prednisolone for doping purposes (systemic and not intra-articular use), it is therefore necessary to know the urinary elimination kinetics of prednisolone and prednisone, as well as the evolution of the concentration ratio between these 2 molecules.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female
* 18-65 years old
* requiring intra-articular injection of prednisolone as part of routine care
* naive to any corticosteroid administration
* requiring a blood biology test as part of routine care and before the infiltration procedure
* For women of childbearing age, negative urine pregnancy test at inclusion
* Affiliated to a social health insurance plan
* Able to understand the protocol and give free, informed and written consent

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient consulting the rheumatology department of the university hospital of Strasbourg (France) for a knee pathology requiring a glucocorticoid infiltration.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Pre-intervention (infiltration)
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Hour24 after intervention
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Hour48 after intervention
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Day7 after intervention
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Day14 after intervention
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Day28 after intervention
  Urinary dosing
Qualitative urinary determination (presence or absence) by LC-MS/MS of the prednisolone/prednisone ratio at specific times | Day42 after intervention
  Urinary dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Laurent MONASSIER, Strasbourg, France